CLINICAL TRIAL: NCT06671821
Title: HRS-7535-202 Follow-up Study: A Long-term Evaluation of Safety, Tolerability, and Efficacy in Obese Subjects (Open-label, Extension Trial)
Brief Title: Long-term Efficacy and Safety of HRS-7535 Tablets in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-202-Extension
Record Dates: First submitted 2024-10-23; First posted 2024-11-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Chronic Weight Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Subjects will receive escalated dose of HRS-7535 or maximum tolerated dose orally
  Interventions: Drug: HRS-7535
- Group B (Experimental): Subjects will receive escalated dose of HRS-7535 or maximum tolerated dose orally
  Interventions: Drug: HRS-7535
- Group C (Experimental): Subjects will receive escalated dose of HRS-7535 or maximum tolerated dose orally
  Interventions: Drug: HRS-7535
- Group D (Experimental): Subjects will receive escalated dose of HRS-7535 or maximum tolerated dose orally
  Interventions: Drug: HRS-7535

INTERVENTIONS:
Drug: HRS-7535 — HRS-7535

SUMMARY:
The Objective of this trial is to evaluate the long-term safety, tolerability, weight loss efficacy and metabolic benefits of HRS-7535 tablets inobesity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-65 years of age at the time of signing informed consent;
2. Subjects who have completed the entire 36-week treatment course of the HRS-7535-202 trial.
3. Subjects who have a full understanding of the trial content, processes, and possible adverse reactions, and are capable and willing to comply with the protocol requirements to complete this study.

Exclusion Criteria:

1. Participants with poor compliance during the 36-week open-label extension treatment of the HRS-7535-202 trial;
2. Pregnant, lactating, planning to conceive during the trial period, or fertile subjects unwilling to take effective contraceptive measures during the trial period.
3. Any other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Event(AE) | During the 32-week open-label extension treatment period

SECONDARY OUTCOMES:
Percentage change in body weight from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment; | from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment;
Proportion of subjects with ≥5%, ≥10%, and ≥15% weight reduction from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment; | from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment;
Changes in weight from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment; | from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment;
Changes in waist circumference from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment; | from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment;
Changes in body mass index (BMI) from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment; | from baseline before HRS-7535 tablet treatment to Week 32 of open-label extension treatment;

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided